CLINICAL TRIAL: NCT04595604
Title: Long Term Effect of Trimodal Prehabilitation Compared to ERAS in Colorectal Cancer Surgery.
Acronym: Prehab_2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Borbala Hospital (Other Government)
Collaborators: Biological Research Centre, Szeged (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ERASvsPrehab_2
Record Dates: First submitted 2020-09-30; First posted 2020-10-20 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer
Keywords: ERAS; prehabilitation; fecal microbata
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Preoperative Exercise; Enhanced Recovery After Surgery

STUDY DESIGN:
Intervention Model Description: Patients planned for elective, curative operations for colorectal cancer will be randomized into two groups: experimental group will take part in a dedicated 4-week multimodal preparation program followed by ERAS preoperative management, while control group will just participate in the ERAS program without specific physical and mental preparation.
  2:1 randomization will be performed for interventional and control arm
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and assessors will be blinded regarding preoperative preparation. Both randomization process and rehabilitation process will be carried out by a trained nurse, physiotherapist and psychotherapist, neither of them will be involved in outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trimodal prehabilitation + ERAS (Experimental): Patients receiving a formal preoperative preparation on:
  Physical status (walking, respiratory training) Nutrition (nutritional supplements) Mental status (weekly groups led by clinical psychologist on anxiety and depression management).
  Each patient will be treated in an ERAS program preoperatively.
  Interventions: Procedure: Trimodal rehabilitation + ERAS
- ERAS + nutritional prehabilitation (Active Comparator): Each patient will be treated in an ERAS program preoperatively. No specific preoperative training will be involved apart from nutritional status assessment and nutritional supplements.
  Interventions: Procedure: ERAS + nutritional prehabilitation

INTERVENTIONS:
Procedure: Trimodal rehabilitation + ERAS — Prehabilitation will cover a range preoperative education and exercises (weekly) on diet, physical activity (daily walking), respiratory training (forced deep inspiration with spirometer device), as well as anxiolytic group psychotherapy.
  Other Names: Prehabilitation
  Arms: Trimodal prehabilitation + ERAS
Procedure: ERAS + nutritional prehabilitation — Enhanced Recovery Program, including preoperative 4 weeks nutritional supplementation.
  Other Names: Enhanced Recovery After Surgery
  Arms: ERAS + nutritional prehabilitation

SUMMARY:
Elective surgery is the most effective treatment option for colorectal cancer, however it has been recognized to be associated with high morbidity and mortality risks.

ERAS (Enhanced Recovery After Surgery) is a preoperative multimodality treatment package, which has been well investigated and proved to be effective in reducing early postoperative morbidity, mortality, length of hospital stay and hospital costs, as well. Still, a good proportion of patients are not suitable for ERAS program, mainly based on lack of compliance and the impaired physical function before surgery.

Trimodal Prehabilitation Program is a recently introduced preoperative preparation (training) program, which addresses improvement of physical, mental and nutritional status of the high risk elective surgery patients.

This study aims to investigate the benefit of all efforts of a 4-6-week preoperative preparation program (Prehabilitation) being added to an established ERAS protocol.

Additionally the effect of trimodal prehabilitation on gut microbiom diversity and its relation to clinical outcome will be analyzed.

DETAILED DESCRIPTION:
Aim:

Colorectal cancer patients with a planned resection are tested if a complex, trimodal rehabilitation program can hold functional and morbidity benefit for them.

In the prospective, randomized (2:1) study control patient group will be the well established and tested ERAS (enhanced recovery after surgery) Program.

Study protocol in details:

First visit: Outpatient Department of Surgery

On both arms:

* History taking (including family history and oncologic history);
* Physical examination

Operation indication, type of procedure and date of procedure agreed; Organizing further investigations, anesthesia; Operative risk assessment ("ACS - surgical risk calculator"); Study patient identifier Nr generated; Nurse-led ERAS/Prehab clinic: randomization

On both arms:

* Randomization (Prehabilitation Program / ERAS Program). 2:1
* Nurse led clinic assessment ("study nurse"):

.i. CaseReportForm (CRF) filled in.

.ii. Patient data (personal data, demographics, history) .iii. Anthropometrics (BMI, MUST, Body fat % measurement). .iv. Mental hygienic status assessment (smoking, alcohol consumption, anxiety, depression, sleeping disorders).

.v. Cardiovascular status (resting HR, RR). .vi. Operative risk assessment (CR-Possum score). .vii. Preoperative counseling (operation type, preparation, pain management, discharge plan).

.viii. Preoperative nutritional planning (education, nutrient prescription). .ix. Alcohol intake and smoking cessation - information given. .x. Stoma education started. . xi. Consent signed, patient workbook handed over. .xii. Respiratory test referral. xiii. Fecal sample collected and stored at -86 C.

Physiotherapy, first visit

Both on control and interventional arms:

* Respiratory function test recorded.
* Physical status tested (6MWD) on a treadmill.

Just on Prehabilitation arm:

* Respiratory training education.
* Respiratory trainer device usage educated.
* Daily activity (walking) planned.

Physiotherapy - second/third/fourth visit (weekly)

Just on Prehabilitation arm:

Previous week activity reviewed as to workbook. Physical assessment: 6MWD, FVC. Next week activity planned. Psychic preparation

Just on Prehabilitation arm:

• Once a week half an hour group relaxation training - regardless of the stage of prehabilitation program.

Admission to the Surgical Ward a day before surgery

Both on control and interventional arm:

* Preoperative assessment:

.i. Anthropometrics (BMI, body fat%). .ii. Cardiovascular stage (resting HR and RR), ECG. .iii. Respiratory function tests. .iv. Physical status (6MWD) .v. Mental status (Hospital Anxiety and Depression Scale (HADS)) assessment. vi. Fecal sample collected and stored at -86 C.

* Preoperative preparation (as to ERAS protocol).
* Postoperative care (ITU, pain management, mobilization, oral nutrition built up, drains early removal, complications recorded (Clavien-Dindo-classification)).
* Stoma education.

Dietary education. On discharge: Quality of Life (QoL) SF36 - (36-Item Short Form Survey from the RAND Medical Outcomes Study).

Postoperative follow up:

Both on control and interventional arms:

• Assessment (8th week post op.):

.i. Anthropometrics (BMI, Body fat %) .ii. Cardiovascular status (resting HR and RR). .iii. Respiratory function tests. .iv. Physical status (6MWD). .v. Fecal sample collected and stored at -86 C.

- Long-term follow-up: 12, 24, 36, 48 and 60 months post operative assessment: Behavioral changes (alcohol abstinence, smoking cessation) Daily physical activity routine assessment. SF36 quality of life assessment Oncological outcome: local recurrence rate, distant recurrence rate, disease free survival, overall survival.

ELIGIBILITY:
Inclusion Criteria:

* patient with histologically proven primary colorectal adenocarcinoma
* any stage of colorectal cancer
* elective operation
* curative intention
* informed consent signed by patient

Exclusion Criteria:

* emergency operation
* palliative operation
* non-colorectal, second malignancy
* pregnancy
* patient not giving consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2022-08-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | 45 days
  Postoperative length of hospital stay in days.
Number of days spent on ICU (Intensive care unit). | 45 days
  Number of days observed on ICU right after operation.
Morbidity (early) classified after Clavien-Dindo. | 7 days (until 8th postoperative day) postoperative
  7-day morbidity will be detailed assessed. Grade 3 or above morbidity rate will be assessed.
Morbidity (long term) classified after Clavien-Dindo. | 30 days (until 31st postoperative day)
  30-day morbidity will be detailed assessed. Grade 3 or above morbidity rate will be assessed.
30-day mortality | 30 days (until 31st postoperative day)
  30-day mortality of each patient will be recorded.
90-day mortality | 90 days (until 91st postoperative day)
  90-day mortality of each patient will be recorded.
Change in preoperative functional status - 6MWD by operation | Measured points: 4 weeks before surgery, on day of hospital admission
  6MWD (6-minute walking distance test)
Change in postoperative functional status - 6MWD by the end of rehabilitation | Measured points: 4 weeks before surgery, 8 weeks after operation
  6MWD (6-minute walking distance test)
Change in preoperative functional status - FVC by operation | Measured points: 4 weeks before surgery, on day of hospital admission
  Measured points: 4 weeks before surgery, on day of hospital admission
Change in preoperative functional status - FVC by the end of rehabilitation | Measured points: 4 weeks before surgery, 8 weeks after operation
  Measured points: 4 weeks before surgery, 8 weeks after operation

SECONDARY OUTCOMES:
Change of alpha- and beta-diversity of fecal microbata | Measured points: 4 weeks before surgery, on day of hospital admission and 8 weeks after surgery
  Fecal microbara diversity will be measured at diagnosis, at the time of operation and 8 weeks after operation. We will assess diversity changes related to the intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- Hungary (2):
  - Department of Surgery, St. Borbala Hospital, Tatabánya
  - St. Borbala Hospital, Tatabánya

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 10 years

REFERENCES:
- [Derived] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub3. PMID 37162250
- [Derived] Molenaar CJ, van Rooijen SJ, Fokkenrood HJ, Roumen RM, Janssen L, Slooter GD. Prehabilitation versus no prehabilitation to improve functional capacity, reduce postoperative complications and improve quality of life in colorectal cancer surgery. Cochrane Database Syst Rev. 2022 May 19;5(5):CD013259. doi: 10.1002/14651858.CD013259.pub2. PMID 35588252